CLINICAL TRIAL: NCT04868994
Title: Contribution of Whole Body Muscle MRI for Early Diagnosis of Amyotrophic Lateral Sclerosis.
Brief Title: Magnetic Imaging for Diagnostic of Amyotrophic Lateral Sclerosis
Acronym: MIDALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/20/0217
Record Dates: First submitted 2021-03-26; First posted 2021-05-03 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis With Dementia
Keywords: Amyotrophic; Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENMG and muscle analyses on whole body muscles MRI. (Experimental): Diffusion of active and chronic muscle denervation will be assessed on ENMG and whole body muscle MRI. The diagnostic category will be determined by revised El Escorial criteria and Awaji criteria
  Interventions: Diagnostic Test: Whole Body MRI and ENMG

INTERVENTIONS:
Diagnostic Test: Whole Body MRI and ENMG — Whole body muscle MRI lasting 30 to 45 min without injection of contrast medium an ENMG

SUMMARY:
Nearly 60% of Amyotrophic Lateral Sclerosis (ALS) patients have a low level of diagnostic certainty (possible, probable) at the time of diagnosis. In the absence of biomarkers, this diagnosis is based, among other things, on the demonstration of the diffusion of signs of denervation by electroneuromyography (ENMG). The objective of this study is to improve the earliness and the level of diagnostic certainty by better demonstrating the diffusion of the denervation process by whole body muscular MRI.

DETAILED DESCRIPTION:
The objective of this study is to show that the combination of ENMG and whole body muscle MRI (WB-MRI) can increase the diagnosis of definite ALS at the onset of the disease For 50 consecutive patients with suspected ALS, the present study will prospectively perform needle electromyography (EMG) and muscle analyses on whole body MRI. The diagnostic category will be determined by revised El Escorial criteria and Awaji criteria. On whole body MRI acquisition, for 83 muscles, will be explored fatty infiltration and atrophy on fat images (chronic denervation) and muscle edema on water images (acute denervation). EMG studies will be performed in at least 10 muscles (tongue, biceps brachii, first dorsalis interosseous, T10 paraspinalis, vastus lateralis, and tibialis anterior). Diagnostic classification according EMG and/ or MRI abnormalities in bulbar and the 3 spinal regions will be compared independently.

ELIGIBILITY:
Inclusion Criteria:

* Consent form signed by the patient
* Patients suspected ALS defined according Awaji Shima criteria (possible, probable, defined)
* Clinical assessment of upper motor neuron involvement
* Electrophysiologic assessment of lower motor neuron involvement

Exclusion Criteria:

* inability to give informed consent
* a contraindication to MRI
* respiratory failure impairing ability to lie flat in the scanner.
* Patient placed under judicial protection or under another protective regime,
* Females who are pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic certainty 1.ENMG according to El Escorial revised criteria using ENMG alone, MRI alone and ENMG+MRI to define denervation diffusion | 1 month
  number of patients classified as possible, probable or certain according to El Escorial criteria using ENMG alone, IMR alone and ENMR+MRI

SECONDARY OUTCOMES:
Define precise topographic and characteristic of muscle involvement in ALS by MRI | 1 month
  number of patients with concordance between ENMG and MRI for the detection of denervation

CONTACTS AND LOCATIONS:
Overall Officials: Pascal CINTAS, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Pascal CINTAS, Toulouse, France